CLINICAL TRIAL: NCT01115244
Title: Dapsone Gel, 5% for Topical Treatment of Dermatitis Herpetiformis
Brief Title: Use of Dapsone Gel, 5% for Treating Dermatitis Herpetiformis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor enrollment and lack of funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100273
Record Dates: First submitted 2010-04-23; First posted 2010-05-04 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Dermatitis Herpetiformis
Keywords: Dermatitis herpetiformis; Dapsone
MeSH Terms: conditions — Dermatitis Herpetiformis | interventions — Dapsone; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapsone gel, 5% (Experimental): ACZONE™ (dapsone) Gel, 5% will be applied to one elbow or knee, randomized at time of enrollment. Application will be topical to the same location twice daily (morning and evening) for six weeks.
  Interventions: Drug: Dapsone gel, 5%
- Not treated (No Intervention): One arm of the patient will be left untreated.

INTERVENTIONS:
Drug: Dapsone gel, 5% — ACZONE™ (dapsone) Gel, 5% will be applied to one elbow or knee, randomized at time of enrollment. Application will be topical to the same location twice daily (morning and evening) for six weeks.
  Other Names: ACZONE™ (dapsone) Gel, 5%
  Arms: Dapsone gel, 5%

SUMMARY:
The primary objective of this study is to evaluate the efficacy of dapsone gel, 5% in the treatment of dermatitis herpetiformis. The primary efficacy end point will be the proportion of patients achieving success based on mean % reduction from baseline in total lesion counts at week six. Success for lesion reduction will be defined as statistically greater mean percent reductions at week six in the dapsone gel-treated extremity compared with the control extremity of each patient.

DETAILED DESCRIPTION:
The study will be a prospective evaluation of dapsone gel, 5% in patients with a clinical diagnosis of dermatitis herpetiformis. Active disease must occur on the patients' bilateral elbows or bilateral knees at the time of study enrollment. Active disease will be defined as five or more papules/pustules/vesicles on an extremity. Randomization of one of the patient's extremities (either one elbow or one knee) to the treatment group will occur at time of enrollment. Randomization will be in the sequence of right side assigned to odd numbered patients and left side assigned to even numbered patients. Thus, the first patient to be enrolled, patient number one, would be randomized to treatment on his or her right side. Depending on the site of active disease, he or she would apply topical dapsone gel, 5% to the right elbow or knee twice daily for the duration of the study.

No blinding of the patients or the PI will occur. The co-investigator will be blinded to whether the photographs presented to him at the end of the study are those of a treated or untreated extremity.

The patients will be screened for study enrollment in a private clinic room within the dermatology clinic at One Hundred Oaks. Patients will be presented with a study summary sheet and a consent form. They will be allowed to ask questions pertaining to the study protocol. Information provided to them will be that found in the study protocol alone. If desired, informed consent can be taken home with the patient to consider, and enrollment can be performed at a later date. In that instance, the patient would be brought back for an additional visit at the time of consent and study enrollment. Study enrollment and first treatment will be performed on the day of study consent. Digital photographs of each elbow or each knee (treatment and control) will be taken on the day of enrollment to serve as a baseline evaluation. The number of lesions (including papules, plaques and vesicles) will be recorded for the treatment and control elbow or knee. Measurements of each lesion will be taken and recorded as well. This data will be written in a chart and stored in the PI's notebook in a locked cabinet in the department of dermatology. Digital photographs will be printed out on the same day as the visit and placed in the notebook as well. Two copies of each photograph will be made. Each photograph will be assigned a letter, A through Z, based on a code for each patient. One copy of each set of photographs will also include the date. No patient identifiable features will be included in the photograph such as the face or eyes. Each photograph will be of the treated or control area only. The code to identify patient photographs will be assigned by the Data and Safety Monitor and kept in a separate locked cabinet. The code will be broken following the blinded evaluation of the photographs by co-investigator.

The patient will be given oral instructions regarding the application of topical dapsone gel, 5% by the PI on the day of enrollment. The PI will apply the first treatment to the randomized extremity during the first clinic visit. The patient will then remain in the treatment room for fifteen minutes to evaluate for any immediate adverse reaction. The PI will remain in the room with the patient. At the end of the fifteen minute evaluation, the patient will be sent home with written instructions for application and a 30gm tube of ACZONE™ (dapsone) Gel, 5%. Patients will apply the study drug to the indicated elbow or knee each morning and evening for the two weeks. They will return to the dermatology clinic in two weeks and be seen in a private clinic room by the PI for a follow up visit. At that time, photographs, lesion counts and measurements will be taken again, just as they were at the initial visit. The patient will be asked to report any adverse events at that time. Patients will be instructed to continue treatment and follow up in two weeks. The same parameters will be evaluated at the four week visit and again at the six week visit, which will be the completion of the study.

Patients will discontinue treatment after six weeks. The co-investigator will be presented will all photograph marked with the patient letter only. He will not know the sequence of the photographs or dates taken. He will then assign a number according to his subjective evaluation of the clinical photographs, while also being blinded to which elbow or knee was treated, right or left. The scores assigned will follow the criteria listed in the investigator's Dermatitis Herpetiformis Assessment Score. The code to the photographs will be broken after the completion of photograph evaluation. Photographs of a set will be matched to those with both letter and date to determine the scores in chronological order.

Six weeks after completion of treatment each patient will be contacted by phone and asked a series of five questions. That will conclude the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years or older
* Clinical diagnosis of dermatitis herpetiformis, as previously diagnosed by the patient's primary dermatologist or diagnosed by agreement of the two investigators
* Active disease at time of enrollment, defined as at least five inflammatory lesions (to include papules, plaques and vesicles) on the bilateral elbows or bilateral knees

Exclusion Criteria:

* Patients taking oral dapsone or those who have taken oral dapsone within four weeks prior to enrollment
* Patients using any other topical treatment for dermatitis herpetiformis at time of enrollment or within the four weeks prior to enrollment
* Patients with known allergy or hypersensitivity to dapsone, sulfa drugs or excipients of the dapsone gel product
* Women will be excluded if pregnant or nursing
* Women of childbearing potential must be practicing an effective method of birth control as determined by the enrolling physician. If oral contraceptives are the method of choice, then the patient must have been on a stable dose for a minimum of 3 months. (This is the same guideline used for women of childbearing potential in previous studies of acne patients.)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University - One Hundred Oaks, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was consented for this study but never returned for the initial study visit and did not receive treatment.
Period: Overall Study
Arm/Group | Dapsone Gel, 5% | Not Treated
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapsone Gel, 5% | Not Treated | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number and Size of All Lesions on the Treated and Untreated Elbows or Knees of Patients With Dermatitis Herpetiformis Who Have One Extremity Treated With Dapsone Gel, 5%
Description: The primary objective is to evaluate the efficacy of dapsone gel, 5% in the treatment of dermatitis herpetiformis. The primary efficacy end point will be the proportion of patients achieving success based on mean % reduction from baseline in total lesion counts at week six. Digital photographs of each elbow or each knee (treatment and control) will be taken. The number and size of lesions will be recorded for the treatment and control elbow or knee. This process will be repeated at each follow up visit.
Time Frame: 6 weeks of treatment
Arm/Group | Dapsone Gel, 5% | Not Treated
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Papules, Plaques and Vesicles on Treated and Untreated Elbows or Knees of Patients Who Have One Extremity Treated With Dapsone Gel, 5%
Description: Lesion types will be counted at recorded at each visit. The mean lesion counts for papules, plaques and vesicles, as well as mean reduction of disease burden from baseline at week six for each of these categories, will be determined.
Time Frame: 6 weeks of treatment
Arm/Group | Dapsone Gel, 5% | Not Treated
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Evaluation of Clinical Photographs and Scoring of Photographs Based on a Modified Global Acne Assessment Score
Description: Photographs of the treated and control extremity of each patient will be presented to the investigator in a blinded manner. Scores will be assigned according to a modified Global Acne Assessment Score. This scoring system has previously been used to evaluate the efficacy of dapsone gel, 5% in the treatment of acne. The designated score is based on disease severity, number of lesions, and type of lesions.
Time Frame: 6 weeks of treatment
Arm/Group | Dapsone Gel, 5% | Not Treated
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dapsone Gel, 5% | Not Treated
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes